CLINICAL TRIAL: NCT03953313
Title: Risk Communication About Post-operative Delirium (POD) and Post-operative Cognitive Dysfunction (POCD)
Status: Completed | Type: Observational
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Claudia Spies, Head of the Department of Anesthesiology and Operative Intensive Care Medicine Berlin (CCM/CVK), Charité - Universitätsmedizin Berlin, Charite University, Berlin, Germany
Other Study IDs: RISKOMMDELIR
Record Dates: First submitted 2019-05-10; First posted 2019-05-16 (Actual); Last update posted 2023-02-02 (Actual); Status verified 2023-02

CONDITIONS: Post-operative Delirium; Post-operative Cognitive Dysfunction
MeSH Terms: conditions — Emergence Delirium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to assess the awareness of post-operative delirium (POD) and post-operative cognitive dysfunction (POCD), their respective risk factors and effective preparation and treatment options in a pre-clinical sample of patients attending a premedication outpatient clinic (Charité - Universitätsmedizin Berlin, Campus Virchow-Klinikum, Berlin, Germany) prior to elective surgery.

The investigators hypothesize that the awareness for POD/POCD as potential risk in consequence of the surgery is very low in patients, and that therefore easy to use measure for prevention are underutilized by patients.

DETAILED DESCRIPTION:
A post-operative delirium is defined as attentional, consciousness and perceptual deficit occurring after and as a consequence of an operation. These deficits are acute and severe, but usually reversible. A post-operative cognitive dysfunction (POCD) is a serious impediment to cognitive functioning, affecting memory, learning, and cognition, again occurring after and as a consequence of an operation. Both delirium and POCD, of which delirium is predictive, have been recognized in medical science as being associated with major cardiac surgery for a while. However, its prevalence after non-cardiac surgery and its links to mortality have only been quantified relatively recently. These studies show that delirium and POCD are very frequent post-operative complications that often go unrecognized. The prevalence across different age groups varies: younger (18-39) adults and older (60+) adults seem to be particularly at risk of developing early POCD (i.e., POCD at hospital discharge) with one study reporting 36.6% of younger and 41,4% of older adults being affected, as compared to the middle-aged (40-59), 30.4% of which were affected. Late POCD (i.e., POCD three months after hospital discharge) was found to be significantly more common in older adults (12.7%) than in the younger or middle aged population (5.7% and 5.6%, respectively). In intensive care settings, delirium is estimated to occur in up to 82% of patients, POCD in up to 41%.

Importantly, delirium as well as POCD are associated with significant negative effects on health: Investigators report a 1-year mortality rate post-discharge of 10.2% for patients with late POCD. Investigators conducted a meta-analysis of post-discharge mortality, institutionalization and dementia amongst elderly patients and found a 38.0% risk of death for patients with delirium by the time of a 2-year follow-up, compared to a control group with 27.5%; a 33.4% probability of institutionalization a year later as compared to 10.7% in the control; and a 62.5% chance of developing dementia up to 4 years later as compared to 8.1% in the control. These differences were independent of confounders such as age, sex, comorbidity, illness severity, and baseline dementia scores. Other studies report prolonged cognitive impairment over 12 months after surgery and significantly higher rates of job loss associated with POCD.

Note that delirium and POCD are complications that can be managed very well. There are relatively simple ways to prevent delirium or recover from it more quickly. Importantly, patients themselves can do a great deal in the way of preparation for an operation and post-operative behavior to significantly reduce their likelihood of getting delirium / POCD or manage it successfully. Yet, most patients are only made aware of the issue, if at all, during their pre-operative anesthetic consultation, usually the evening before the operation - too late to put many of the important preparatory behaviours into place. Importantly, there is no direct communication channel between general practitioners, who refer the patient, and clinical anesthesiologists who deal with delirium / POCD management. Thus, risk factors for as well as incidence of delirium / POCD after surgeries are likely not passed between these important actors in the health system.

Given its high prevalence and serious impact on mental health, physical health, and socio-economic factors, it is imperative that patients and general practitioners alike are aware of delirium / POCD as well as how to recognize it, how to best prepare for an operation in order to reduce its chance of occurrence, and how to behave in case post-operative delirium or POCD has developed. To the knowledge of the investigators, this is the first study to date assessing the awareness of delirium / POCD, their respective risk factors and effective preparation and treatment options in a pre-clinical sample of the general population. Goal of the study is to assess and quantify the current communication deficit in the healthcare system and thus build up pressure to improve it.

ELIGIBILITY:
Inclusion Criteria:

* male or female patients attending the premedication outpatient clinic Charité University Medicine, CVK, Berlin, Germany in order to attend a (non-cardiac) elective surgery
* 18 years or older

Exclusion Criteria:

* Refusal by the patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male or female adult patients attending the premedication outpatient clinic Charité University Medicine, CVK, Berlin, Germany in order to attend a (non-cardiac) elective surgery
Sampling Method: Probability Sample
Enrollment: 223 (Actual)
Dates: Start 2021-05-03 (Actual); Primary Completion 2021-12-19 (Actual); Study Completion 2021-12-19 (Actual)

PRIMARY OUTCOMES:
Awareness of POD specifically as post-operative complications (Q2) | Prior to elective surgery
  A questionnaire is used to assess this outcome measure awareness of POD as post-operative complications. Response to Question: "A possible complication of an operation can be states of confusion, forgetfulness or problems with thinking / speaking, which usually subside within a few hours or days. This is termed "post-operative delirium. Have you ever heard of this complication?": Yes/No
Awareness of POCD specifically as post-operative complications (Q3) | Prior to elective surgery
  A questionnaire is used to assess this outcome measure awareness of POCD as post-operative complications. Response to Question: "A possible complication of an operation can be a long-term disruption of thinking and a lower mental capacity, which may last up to several months or even years. This is termed "post-operative cognitive dysfunction". Have you ever heard of this complication?": Yes/No

SECONDARY OUTCOMES:
Awareness of post-operative complications (Q1) | Prior to elective surgery
  A questionnaire is used to assess this outcome measure awareness of post-operative complications. Response to question "Which of the following symptoms (pain, wound infection, damage to teeth, sepsis, forgetfulness, loss of orientation, thrombosis, attention deficits, nausea, stroke, heart attack, problems with healing of the wound) do you think are possible immediate consequences of an elective operation (e.g. as opposed to an emergency operation)?": Yes/No
Estimation about prevalence of POD after elective, non-emergency surgeries (Q4) | Prior to elective surgery
  Estimation about prevalence of POD. Answer to Question: "Please estimate, after how many of 1000 operations (no emergencies), patients suffer from a post-operative delirium?": Number range in 1000
Estimation about prevalence of POCD after elective, non-emergency surgeries (Q5) | Prior to elective surgery
  Estimation about prevalence of POCD. Answer to Question: "Please estimate, after how many of 1000 operations (no emergencies), patients suffer from a POCD?": Number range in 1000
Estimation about personal risk of developing POD (Q6) | Prior to elective surgery
  A questionnaire is used to assess this outcome measure patients estimation about personal risk of experiencing postoperative delirium after elective surgery. Answer to Question:" Please estimate your personal risk of suffering a post-operative delirium in percentage points!"
Estimation about personal risk of developing POCD (Q7) | Prior to elective surgery
  A questionnaire is used to assess this outcome measure patients estimation about personal risk of experiencing POCD after elective surgery. Answer to Question: "Please estimate your personal risk of suffering from a post-operative cognitive dysfunction three months after the operation in percentage points!"
Knowledge about preventive measures to reduce likelihood of developing delirium / POCD (Q8) | Prior to elective surgery
  A questionnaire is used to assess this outcome measure the knowledge about preventive measures to reduce likelihood of developing pOD / POCD. Answer to question:" Which of the pre-operative measures (bodily hygiene, taking sedatives or anti-depressants, prepare in a calm, quiet environment for the operation, avoid distractions, drink water until 2 hours prior to the operation, a good night's sleep, avoiding contact with animals (e.g., pets), a protein-rich diet, keeping a diary) do you consider effective in preventing a post-operative Delirium or cognitive dysfunction?": Yes/No
Knowledge about ways to recover from POD / POCD (Q9) | Prior to elective surgery
  A questionnaire is used to assess this outcome measure knowledge about ways to recover from POD / POCD. Answer to Question: " If a delirium or post-operative cognitive deficit occurs, which of the following measures (go home as quickly as possible, avoid distractions or disturbances, pain management with medications in the hospital, mental effort (e.g., playing video games, crossword puzzles, etc.), eating healthy food, taking physiotherapy classes, avoiding daylight, request a single-room in Hospital) do you think is most effective in order to recover from it quickly after the operation?: Yes/No
Patient-specific risk factors of developing POD / POCD (Q10a) | Prior to elective surgery
  A questionnaire is used to assess this outcome measure patient-specific risk factors of developing POD / POCD. Answer to Questions: "Your gender?": male or female
Patient-specific risk factors of developing POD / POCD (Q10b) | Prior to elective surgery
  A questionnaire is used to assess this outcome measure patient-specific risk factors of developing POD / POCD. Answer to Questions: "Your age in years?"
Patient-specific risk factors of developing POD / POCD (Q10c) | Prior to elective surgery
  A questionnaire is used to assess this outcome measure patient-specific risk factors of developing POD / POCD. Answer to Questions: "How many different types of medication to you currently take on a regular basis (please also include medications you do not take due to illness or infection, such as regular intake of aspirin)?": 0,1,2,3,4,5 or more
Patient-specific risk factors of developing POD / POCD (Q10d) | Prior to elective surgery
  A questionnaire is used to assess this outcome measure patient-specific risk factors of developing POD / POCD. Answer to Questions: "In the last 10 years, how often have you been operated on?":0,1,2,3,4,5 or more?
Patient-specific risk factors of developing POD / POCD (Q10e) | Prior to elective surgery
  A questionnaire is used to assess this outcome measure patient-specific risk factors of developing POD / POCD. Answer to Questions: "Have you been diagnosed with one or more of the following illnesses / conditions? -Dementia,-Depression,- Physical Disability,- Seeing or Hearing Problems,-Underweight,- Chronic liver or kidney Damage,-Diabetes,-HIV,-Infection,-Alcohol or drug abuse,-Stroke,-Cardio-vascular Problems?"
Knowledge of the healthcare system (Q10f) | Prior to elective surgery
  A questionnaire is used to assess this outcome measure knowledge of the healthcare System. Answer to Question: "Are you employed in a medical or nursing profession?" Yes/No
Information transfer in healthcare system (Q11) | Prior to elective surgery
  A questionnaire is used to assess this outcome measure information transfer in healthcare System. Answer to Question: "If you have had an elective operation before, has your General practitioner or other medical professional made you aware of the possibility of postoperative delirium or cognitive dysfunction as well as measure of prevention, optimal preparation and treatment?": Yes/No
(Health) behavioral consequences of POD / POCD knowledge (Q12) | Prior to elective surgery
  A questionnaire is used to assess this outcome measure (Health) behavioral consequences of POD / POCD Knowledge. Answer to question: "If you have had an elective operation before, would this information about POD / POCD have influenced your decision to do the operation (i.e., would you have not done it in this case)?": Yes/No
(Health) behavioral consequences of POD / POCD knowledge (Q13) | Prior to elective surgery
  A questionnaire is used to assess this outcome measure (Health) behavioral consequences of POD / POCD Knowledge. Answer to question: "Will these informations about POD / POCD influence your future decisions of whether to do an elective surgery or not?": Yes/No
(Health) behavioral consequences of POD / POCD knowledge (Q14) | Prior to elective surgery
  A questionnaire is used to assess this outcome measure (Health) behavioral consequences of POD / POCD Knowledge. Answer to Question: "Will these informations about POD / POCD influence the way in which you will prepare for elective operations in the future?": Yes/No

CONTACTS AND LOCATIONS:
Overall Officials: Claudia Spies, MD. Prof., Study Director — Charite University, Berlin, Germany
Locations (1):
- Department of Anesthesiology and Operative Intensive Care Medicine Berlin (CCM/CVK), Charité - Universitätsmedizin Berlin, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No